CLINICAL TRIAL: NCT03857386
Title: Comparison of The Effects of Pectoral Nerve Block and Local Infiltration Anesthesia on Postoperative Analgesia for Breast Reduction Surgery
Brief Title: Efficacy of Pectoral Nerve Block for Breast Reduction Surgery
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Arzu Karaveli, study director, Antalya Training and Research Hospital
Other Study IDs: 10/09
Record Dates: First submitted 2018-12-18; First posted 2019-02-28 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Nerve Blocks; Breast Surgery; Postoperative Pain
Keywords: pectoral nerve block (PECS block); breast reduction surgery; ultrasonography; postoperative pain; VAS score
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Conduction; Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PECS group: Preoperative bilateral PECS I + PECS II Pecs block performed by anaesthetist using ultrasound guidance in plane approach
  Interventions: Procedure: PECS group
- Control group: Bilateral local anesthesia infiltration Local infiltration anesthesia performed by surgeon during the operation
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: PECS group — Pecs block performed using ultrasound guidance
  Other Names: Regional anesthesia in breast surgery
  Groups: PECS group
Procedure: Control group — Local infiltration anesthesia performed during the operation
  Other Names: Regional anesthesia in breast surgery
  Groups: Control group

SUMMARY:
The purpose of the study is to evaluate the efficacy of PECS block applied to patients undergoing bilateral breast reduction surgery on postoperative analgesia compared to local infiltration anesthesia.

DETAILED DESCRIPTION:
Pectoral nerve block (PECS block) has been developed as an alternative to thoracic paravertebral and/or thoracic epidural blocks in recent years. It is frequently applied for postoperative analgesia especially in breast cancer surgery and subpectoral breast prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) I-II
* body mass index (BMI) ≤40 kg/m2
* elective bilateral breast reduction surgery

Exclusion Criteria:

* declining to give written informed consent
* ASA III and above
* under 18 years of age or over 65 years of age
* history of allergy against to the local anesthetics,
* controendication of peripheral block or local anesthetic infiltration (local infection, coagulopathy, etc.)
* history of breast surgery
* treatment due to psychiatric disorder
* history of treatment for a chronic pain
* history of nerve blocks in order to treat postoperative pain

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included patients with ASA I-II, 18-65 years old, with a BMI ≤ 40 kg/m2 and undergoing elective breast reduction operation under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
postoperative visual analog scale (VAS) score | postoperative 0, 1, 3, 6, 9, and 12 hours
  Postoperative pain assessment will be performed using the VAS score (VAS 0 = no pain, VAS 10 = most severe pain possible). The VAS scores will be recorded at postoperative 0, 1, 3, 6, 9, and 12 hours.

SECONDARY OUTCOMES:
analgesia consumption | 12 hours
  postoperative
length of hospital | 4 days
  recorded at the following time after surgery
analgesia consumption | during the surgery
  intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Karaveli, Principal Investigator — Netherlands: Ministry of Health, Welfare and Sports
Locations (1):
- Antalya Training and Research Hospital, Department of Anesthesiology and Reanimation, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099